CLINICAL TRIAL: NCT05461937
Title: A Feasibility Randomised-Controlled Trial of Two Online Psychological Interventions for Stroke Survivors
Brief Title: Feasibility Randomised-Controlled Trial of Online Stroke Interventions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of East Anglia (Other)
Responsible Party: Principal Investigator, Catherine Ford, Clinical Associate Professor in Clinical Psychology, University of East Anglia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRAS305848
Record Dates: First submitted 2022-06-30; First posted 2022-07-18 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Stroke
Keywords: Stroke; Executive Functions; Goal Management; Problem-Solving; Psychoeducation; Telerehabilitation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 'Getting things done after stroke' - an online executive function intervention (Experimental)
  Interventions: Behavioral: Getting things done after stroke
- Stroke psychoeducation (Active Comparator)
  Interventions: Behavioral: Stroke psychoeducation

INTERVENTIONS:
Behavioral: Getting things done after stroke — A two-session, online rehabilitation intervention focussing on cognitive executive functions supplemented with weekly homework tasks.
  Arms: 'Getting things done after stroke' - an online executive function intervention
Behavioral: Stroke psychoeducation — A two-session, online stroke psycho-education intervention supplemented with weekly homework tasks.
  Arms: Stroke psychoeducation

SUMMARY:
Many people have difficulties organising their behaviour and problem-solving (also known as executive function difficulties) after stroke. This can have serious, wide-ranging consequences for wellbeing and ability to regain independence. Currently, access to psychological interventions after stroke varies and there is not enough evidence to recommend a specific intervention for executive function difficulties after stroke. A short intervention was designed to help with executive function difficulties by making it easier to set goals and achieve them after stroke. The intervention is designed for online delivery to make it accessible to as many stroke survivors as possible. The present trial aims to investigate the acceptability and feasibility of a single blinded randomized controlled trial of this online executive function intervention (active intervention) compared to an online stroke psychoeducation intervention (control intervention).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of stroke
* ≥ 18 years of age
* Capacitous consent to participate
* Access to a computer / tablet, the internet, and an email address

Exclusion Criteria:

* Another significant mental or physical health condition
* Current involvement in another research trial
* Severe depression (over 20 on PHQ-9)
* Not able to read or understand English
* Visual, auditory or motor difficulties of a severity that limit the ability to attend to the content of the interventions, read the Participant Information Sheet or complete the consent form and outcome measures
* Not registered with a GP or unwilling to provide GP information (for reporting suicidal ideation concerns

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2022-06-10 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Recruitment Rate | Through study completion, approximately 15 months.
  Rate of participants recruited into the trial amongst all participants screened
Exclusion Rate | Through study completion, an average of 15 months.
  Rate of participants excluded from participating amongst all participants screened
Attrition Rate | Through study completion, an average of 15 months.
  Rate of participants and data lost
Follow-up rate | Through study completion, an average of 15 months.
  Rate of participants included at 1-month follow-up
Time required to collect and analyze data | Through study completion, an average of 15 months.
  Time required for data collection per participant and final analysis
Questionnaire reminders | Through study completion, an average of 15 months.
  Number of questionnaire reminders sent and time taken per participant
Support to complete questionnaires | Through study completion, an average of 15 months.
  Number of participants requiring support to complete questionnaires and time taken per participant

SECONDARY OUTCOMES:
The stroke self-efficacy scale (SSES; Jones et al., 2008) | Baseline, post-intervention and at 1-month follow-up.
  A 13-item measure of confidence for functional performance and aspects of self-management relevant post-stroke. Respondents are asked to rate their confidence that they can do various tasks that may have been difficult after having a stroke using a 4-point scale (0=not at all confident, 3=very confident).
The Short Warwick-Edinburgh Mental Wellbeing Scale (SWEMWBS, Tennant et al., 2007) | Baseline, post-intervention and at 1-month follow-up.
  A 7-item questionnaire covering subjective wellbeing and psychological functioning. Respondents are asked to rate each of the items on a scale of 1 to 5 on the basis of how often they had experienced a symptom over the last 2 weeks (1=none of the time, 2=rarely, 3=some of the time, 4= often, 5=all of the time).
Revised Dysexecutive Questionnaire (DEX-R; Simblett, Ring & Bateman, 2016) | Baseline, post-intervention and at 1-month follow-up.
  A tool for measuring everyday problems experienced with the dysexecutive syndrome. It consists of 37 items and respondents are asked to rate how often they experience difficulties related to executive functioning (0=never, 1=occasionally, 2=sometimes, 3=fairly often, 4=very often).
The Patient Health Questionnaire-9 (PHQ-9) | Screening
  A self-report measure of depression consisting of nine items matching the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) criteria of major depression. Respondents are asked to rate each of the items on a scale of 0 to 3 on the basis of how much a symptom has bothered them over the last 2 weeks (0=not at all, 1=several days, 2=more than half the days, 3=nearly every day).
The ICECAP-A (ICEpop CAPability measure for Adults; Al-Janabi, Flynn & Coast, 2012) | Baseline, post-intervention and at 1-month follow-up.
  A measure of capability for the general adult (18+) population for use in economic evaluation. It comprises five attributes (attachment, stability, achievement, enjoyment, and autonomy). Each capability item has four levels of responses.
Feedback survey | Post-intervention.
  A mixture of open-ended (free text response) and closed (Likert type response) questions to assess trial and intervention acceptability.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine EL Ford, PhD, Study Director — University of East Anglia
Locations (1):
- University of East Anglia, Norwich, Norfolk, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ene CG, Gracey F, Ford C. A feasibility randomized-controlled trial of an executive functioning telerehabilitation intervention for stroke survivors. Brain Inj. 2025;39(9):772-783. doi: 10.1080/02699052.2025.2483449. Epub 2025 Mar 27. PMID 40143638